CLINICAL TRIAL: NCT05231772
Title: The Effect of Probiotics on Hemodynamic Changes and Complications of Cirrhosis
Brief Title: Probiotics and Hemodynamic Changes in Cirrhosis
Acronym: PrBHCCir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2533644
Record Dates: First submitted 2022-01-27; First posted 2022-02-09 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-01

CONDITIONS: Cirrhosis
Keywords: gut-liver axis; microbiota; microbiome; liver; cirrhosis; hemodynamics
MeSH Terms: conditions — Fibrosis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Patients in the Test arm will receive Saccharomyces boulardii (Saccharomyces), (Enterol), Biocodex Ltd, France, registration number LP-000622 from 21.09.2011 at a dose of 250 mg 2 times a day for 3 months.
  Interventions: Drug: Saccharomyces Boulardii Probiotic Supplement
- Placebo (Placebo Comparator): Patients in the Placebo arm will receive the placebo at a dose of 250 mg 2 times a day for 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saccharomyces Boulardii Probiotic Supplement — Probiotic yeast
  Other Names: Probiotics; Enterol
  Arms: Probiotics
Drug: Placebo — Placebo
  Other Names: No other name
  Arms: Placebo

SUMMARY:
This is a single-center blinded randomized interventional placebo-controlled study of the effect of probiotics on hemodynamic parameters and liver function in cirrhosis.

DETAILED DESCRIPTION:
Forty patients with Child-Pugh class B and C cirrhosis will be randomized in a 1.5:1 ratio to test and control arms. Patients in the test arm will receive probiotic Saccharomyces boulardii (A07FA02 - Saccharomyces (Enterol) Biocodex Ltd, France, registration number LP-000622 from 21.09.2011) for 3 months, patients in the control arm will receive placebo for 3 months. All patients also will receive standard treatment: spironolactone 100 mg/day in ascites and carvedilol 12.5 mg/day in esophageal varices. The patients will be blinded. At inclusion and after 3 months after starting of probiotic/placebo treatment, systemic hemodynamics parameters (cardiac output and systemic vascular resistance), liver function (serum albumin and total bilirubin level, international normalized ratio, presence and degree of ascites or hepatic encephalopathy), the gut microbiome, biomarkers of bacterial translocation (presepsin, lipopolysaccharide), intestinal permeability (claudin 3), systemic inflammation (tumor necrosis factor alpha ) and endothelial dysfunction (nitrites, endothelin) will be assessed. After the end of the study, an interim analysis of the effect of the probiotic on aforementioned systemic hemodynamics and liver function indicators will be carried out. If there is a positive effect, a full analysis of all the aforementioned factors contributing to its development will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis
* Child-Pugh class B or C;
* Age between 18 and 70 years;
* Signed informed consent.

Exclusion Criteria:

* Use of lactulose, lactitol, or other prebiotics, probiotics, antibiotics, or metformin in the past 6 weeks before inclusion;
* Alcohol consumption in the past 6 weeks before inclusion;
* Inflammatory bowel disease;
* Cancer;
* Prematurely discontinuation of the consumption of tested probiotic/placebo;
* Started taking antibiotics, other probiotics, or prebiotics during the follow-up period;
* Refusal to participate during the follow-up period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
the change in cardiac output | at inclusion and 3 months after the start of the study
  Transthoracic echocardiography (with Acuson S2000 by Siemens Ltd, USA, registration number 2017/6109 from 24.07.2018) according to the guidelines of the American Society of Echocardiography (published in 2015) with a simultaneous assessment of blood pressure (with semi-automatic tonometer UA-604 by AND Ltd, Japan, registration number 2011/09642 from 10.10.2018) and heart rate will be performed to assess systemic hemodynamics. Cardiac output will be calculated as (stroke volume) × (heart rate).
the change in number of points on the Child-Pugh scale | at inclusion and 3 months after the start of the study
  The scale assesses the degree of hyperbilirubinemia (1 point - serum total bilirubin level is less than 2 mg / dl, 2 points - 2-3 mg / dl, 3 points - above 3 mg / dl), hypoalbuminemia (1 point - serum albumin level above 35 g / l, 2 points - 28-35 g / l, 3 points - less than 28 g / l), hypocoagulation (1 point - international normalized ratio less than 1.7, 2 points - 1.7-2.3, 3 points - above 2.3) degree of ascites (1 points - no ascites, 2 points - ascites detected only with ultrasound, 3 points - large ascites visible to the eyes) of hepatic encephalopathy (1 point - no hepatic encephalopathy; 2 points - hepatic encephalopathy without severe manifestations (stupor or coma); 3 points - severe hepatic encephalopathy (stupor or coma)).

SECONDARY OUTCOMES:
the change in the serum albumin level | at inclusion and 3 months after the start of the study
  venous blood will be take on an empty stomach at 7-9 am without any special preparation
the change in the serum total bilirubin level | at inclusion and 3 months after the start of the study
  venous blood will be take on an empty stomach at 7-9 am without any special preparation
the change in the international normalized ratio | at inclusion and 3 months after the start of the study
  venous blood will be take on an empty stomach at 7-9 am without any special preparation
the change in the serum C-reactive protein level | at inclusion and 3 months after the start of the study
  venous blood will be take on an empty stomach at 7-9 am without any special preparation
the change in systemic vascular resistance | at inclusion and 3 months after the start of the study
  systemic vascular resistance will be calculated as mean arterial pressure/cardiac output
the change in the degree of hepatic encephalopathy | at inclusion and 3 months after the start of the study
  0 - no hepatic encephalopathy, 1 - minimal hepatic encephalopathy (normal neurological status but abnormal number connection test), 2 - overt hepatic encephalopathy (abnormal neurological status)
the change in the degree of ascites | at inclusion and 3 months after the start of the study
  0 points - no ascites, 1 points - ascites detected only with ultrasound, 2 points - ascites detected with the shifting dullness method; 3 point - gross refractory ascites.
the change in the presence of small intestinal bacterial overgrowth | at inclusion and 3 months after the start of the study
  lactulose hydrogene breath test with Gastro+Gastrolyzer (by Bedfont Ltd, the United kingdom, registration number 2010/06253 from 17.09.2020) in accordance with the North American Consensus: the presence of small intestinal bacterial overgrowth is considered when there was an increase in breath hydrogen of at least 20 ppm above the baseline value within 90 minutes after taking 10 ml of lactulose dissolved in 200 ml of water.
the change in the serum presepsin level | at inclusion and 3 months after the start of the study
  venous blood will be take on an empty stomach at 7-9 am without any special preparation
the change in the serum lipopolysaccharide level | at inclusion and 3 months after the start of the study
  venous blood will be take on an empty stomach at 7-9 am without any special preparation
the change in the serum claudin 3 level | at inclusion and 3 months after the start of the study
  venous blood will be take on an empty stomach at 7-9 am without any special preparation
the change in the serum tumor necrosis factor alpha level | at inclusion and 3 months after the start of the study
  venous blood will be take on an empty stomach at 7-9 am without any special preparation
the change in the serum nitrites level | at inclusion and 3 months after the start of the study
  venous blood will be take on an empty stomach at 7-9 am without any special preparation
the change in the serum big endothelin level | at inclusion and 3 months after the start of the study
  venous blood will take on an empty stomach at 7-9 am without any special preparation

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Ivashkin, Prof., Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- Clinic for Internal Diseases, Gastroenterology and Hepatology at Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Data disclosure is not permitted by the Local Ethics Committee of I.M. Sechenov First Moscow State Medical University. For more information about the study, you need to contact the principal investigator.

REFERENCES:
- [Background] Maslennikov R, Ivashkin V, Efremova I, Poluektova E, Shirokova E. Gut-liver axis in cirrhosis: Are hemodynamic changes a missing link? World J Clin Cases. 2021 Nov 6;9(31):9320-9332. doi: 10.12998/wjcc.v9.i31.9320. PMID 34877269
- [Background] Maslennikov R, Ivashkin V, Efremova I, Alieva A, Kashuh E, Tsvetaeva E, Poluektova E, Shirokova E, Ivashkin K. Gut dysbiosis is associated with poorer long-term prognosis in cirrhosis. World J Hepatol. 2021 May 27;13(5):557-570. doi: 10.4254/wjh.v13.i5.557. PMID 34131470
- [Background] Maslennikov R, Ivashkin V, Efremova I, Poluektova E, Shirokova E. Probiotics in hepatology: An update. World J Hepatol. 2021 Sep 27;13(9):1154-1166. doi: 10.4254/wjh.v13.i9.1154. PMID 34630882
- [Background] Ivashkin V, Fomin V, Moiseev S, Brovko M, Maslennikov R, Ulyanin A, Sholomova V, Vasilyeva M, Trush E, Shifrin O, Poluektova E. Efficacy of a Probiotic Consisting of Lacticaseibacillus rhamnosus PDV 1705, Bifidobacterium bifidum PDV 0903, Bifidobacterium longum subsp. infantis PDV 1911, and Bifidobacterium longum subsp. longum PDV 2301 in the Treatment of Hospitalized Patients with COVID-19: a Randomized Controlled Trial. Probiotics Antimicrob Proteins. 2023 Jun;15(3):460-468. doi: 10.1007/s12602-021-09858-5. Epub 2021 Oct 13. PMID 34643888